CLINICAL TRIAL: NCT07171138
Title: Pressure Injury Risk Related to Positioning and Positioning Devices in Burn Patients
Brief Title: This Study Will Use Real-time Pressure Mapping Technology to Determine Which Positioning Strategies and Devices Exert the Least Amount of Pressure on Peri-operative Burn Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 6758
Record Dates: First submitted 2025-08-26; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Hospital Acquired Pressure Injury
MeSH Terms: interventions — Patient Positioning

STUDY DESIGN:
Intervention Model Description: Pre/post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAPI incidence post-implementation of optimal positioning (Active Comparator): Compare HAPI incidence post-implementation of positioning that produced the least pressure with retrospective pre-intervention HAPI incidence
  Interventions: Device: Positioning and positioning devices

INTERVENTIONS:
Device: Positioning and positioning devices — Different positioning strategies and positional devices. Measurement of skin interface pressure at key anatomical pressure points (occiput, elbows, sacrum, heels) under different patient positioning strategies and positional devices.
  The positions that produce the least amount of pressure are identified and will be implemented and compared with pre-intervention hospital acquired pressure injuries (HAPI)
  Other Names: X-sensor pressure mapping mat for determining positions of least amount of pressure

SUMMARY:
Burn patients are especially vulnerable to developing hospital-acquired pressure sores. The goal of this study is to determine which positions and positioning devices exert the least amount of pressure on problem areas such as the heels, the tailbone, the elbow and the back of the head.

With the use of a pressure mapping device, it will allow the investigators to:

1. Identify patients at the highest risk of developing pressure injuries related to positioning/devices.
2. Use the findings to create positioning/device guidelines

By optimizing positioning strategies, the investigators aim to enhance patient comfort, prevent complications, and ultimately improve the overall quality of care for burn patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18 years of age or greater)
* burns of any size
* pre and post-operative patients

Exclusion Criteria:

* pediatric burn patients
* patients with pre-existing (pre-admission) pressure injuries
* patients unable to provide informed consent or decline consent
* patients with large burns that are not expected to survive past 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Measurement of pressure according to pressure mapping system/device (x-sensor) | 1 year
  Using a pressure mapping device, determine which positions and positioning devices create the most/least amount of pressure at known pressure points (occiput, elbows, sacrum, and heels).

SECONDARY OUTCOMES:
Compare HAPI incidence post-implementation of optimal positioning | 1 year
  Compare HAPI incidence post-implementation of positioning that produced the least pressure with retrospective pre-intervention HAPI incidence.

IPD SHARING:
Plan to Share IPD: No